CLINICAL TRIAL: NCT00646750
Title: Autologous Transplantation of Haematopoietic Stem Cells With Conditioning Including Zevalin + BEAM to Patients Suffering From Refractory Large B-cell Diffuse Lymphom
Brief Title: Transplantation With Ybritumomab Tiuxetan (Zevalin) Plus BEAM Regimen in Patients With Refractory Large B-cell Difusse Lymphom
Acronym: Z-BEAM LDGGB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Español de Linfomas y Transplante Autólogo de Médula Ósea (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GELTAMO-Z-BEAM LDGGB; EudraCT No.: 2007-003198 - 22
Record Dates: First submitted 2008-03-17; First posted 2008-03-28 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-02

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: Z-BEAM; Autologous; Lymphoma; GELTAMO
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma | interventions — ibritumomab tiuxetan; Rituximab; Carmustine; Etoposide; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): BEAM preceded by Ybritumomab Tiuxetan (Zevalin)
  Interventions: Drug: Ybritumomab Tiuxetan (Zevalin); Rituximab; BEAM (BCNU, ARAC, VP16 and Melphalan)

INTERVENTIONS:
Drug: Ybritumomab Tiuxetan (Zevalin); Rituximab; BEAM (BCNU, ARAC, VP16 and Melphalan) — Day -21: rituximab. 250 mg/m2 iv
  Day -14: rituximab. 250 mg/m2 plus Ybritumomab Tiuxetan (Zevalin)(0.4 mCi/kg maximum dose 32 mCi).
  Days -6 to -1: BEAM regimen as follows BCNU: 300 mg/m2 over 2 hours, day -6. ARAC: 200 mg/m2/12 hours over 12 hours, days -5 through -2. VP16: 200 mg/m2/day over 2 hours, days -5 through -2. Melphalan: 140 mg/m2/day over 15 minutes, day -1.
  Other Names: Ybritumomab Tiuxetan (Zevalin); Rituximab (Mabthera)

SUMMARY:
To evaluate the efficacy (complete response rate) of Ybritumomab Tiuxetan (Zevalin) administration in the conditioning treatment of patients with refractory large B-cell diffuse lymphoma submitted to autologous transplantation of peripheral blood haematopoietic stem cells.

ELIGIBILITY:
Inclusion Criteria:

1. Give their written informed consent.
2. Abide by at least one of the following conditions:

   * Obtain no partial response after first-line chemotherapy including anthracyclines + rituximab (R-CHOP, R-MegaCHOP, R-EPOCH or the like), or else
   * Absence of partial response after having received salvage (post-induction) chemotherapy including R-IFE, R-ESHAP, R-ICE or the like.
   * Patients on first recidivation who do not attain partial remission after salvage chemotherapy.
   * Patients with transformed lymphoma, on first partial remission (No CR).
3. Stable disease at the time of transplantation.
4. Age ≥ 18 but ≤ 70.
5. Life expectancy of greater than three months.

Additionally, to be able to undergo haematopoietic stem cell transplantation, all patients should satisfy the requirements of routine clinical practice, i.e.:

1. Performance status (ECOG) < 3.
2. FEV1, DLCO and FVC ≥ 50% of the normal theoretical values.
3. Ventricular ejection fraction (through echocardiography or isotope ventriculography) ≥ 50%.
4. Total bilirubin and transaminases < 3 times the normal maximum value, except if attributable to the underlying disease.
5. Creatinine < 2 times the maximum normal value, and creatinine clearance > 40 ml/min, except if attributable to the underlying disease.
6. Absence of symptomatic heart disease, cirrhosis or active B or C virus hepatitis.
7. HIV negative.

Exclusion Criteria:

1. Impossibility of collecting, via apheresis, a number of CD34+ cells ≥ 2 x 106/kg.
2. Known hypersensitivity to mouse proteins.
3. Involvement of CNS by lymphoma.
4. Progressive lymphoma during the month prior to the date of transplantation.
5. Previous radioimmunotherapy.
6. Previous autologous transplantation of haematopoietic stem cells.
7. Pregnant or breastfeeding women, or adults of childbearing age who are not using an effective contraceptive method.
8. Being submitted to treatment in a clinical trial for 30 days prior to entry in this trial.
9. Active psychiatric disease, including addiction disorders.
10. Existence of active not-haematopoietic neoplasia, with the exception of cutaneous basal carcinoma or cervix intraepithelial carcinoma.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-01; Primary Completion 2010-02 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Disease clinical response to treatment - complete response rate. | Pre-transplantation; post-transplantation (one week following Ybritumomab Tiuxetan (Zevalin) administration); And three months post-transplantation

SECONDARY OUTCOMES:
Haematopoietic and extra-haematopoietic toxicity of the Ybritumomab Tiuxetan (Zevalin) plus BEAM regimen. | 36 months
Overall response rate (complete + partial response) | 36 month
Progression-free-survival | 36 month
Overall survival | 96 months
Post-transplantation haematological and immunological reconstitution | Until post-transplantation day +100

CONTACTS AND LOCATIONS:
Overall Officials: Javier Briones, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Dolores Caballero, MD, Principal Investigator — Hospital Clínico Universitario de Salamanca
Locations (18):
- Spain (18):
  - Hospital Universitario de Alicante, Alicante, Alicante
  - H. de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Instituto Catalán de Oncología,, Barcelona, Barcelona
  - H.Universitario de Canarias, Santa Cruz de Tenerife, Canary Islands
  - H.U. Marqués de Valdecilla, Santander, Cantabria
  - H. Reina Sofía, Córdoba, Córdoba
  - Clínica Puerta de Hierro,, Madrid, Madrid
  - H.U. 12 de Octubre,, Madrid, Madrid
  - H.U. Gregorio Marañón,, Madrid, Madrid
  - H.U. La Paz, Madrid, Madrid
  - H.U. La Princesa, Madrid, Madrid
  - M.D. Anderson Internacional, Madrid, Madrid
  - H. Morales Messeguer, Murcia, Murcia
  - H.U. Virgen de la Arrixaca, Murcia, Murcia
  - Clínica Universitaria de Navarra, Pamplona, Navarre
  - H.U. Central de Asturias, Oviedo, Oviedo, Principality of Asturias
  - H. Clínico Universitario de Salamanca, Salamanca, Salamanca
  - H.U. La Fe, Valencia, Valencia